CLINICAL TRIAL: NCT00424216
Title: Direct Current Brain Polarization of Bilateral Prefrontal Cortex
Brief Title: Direct Current Brain Polarization of the Frontal Lobes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 070066; 07-N-0066
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-12-23

CONDITIONS: Healthy
Keywords: Mood; Emotion; Judgment; Cortex; Brain Stimulation; Healthy Volunteer; HV

INTERVENTIONS:
Procedure: DC Polarization

SUMMARY:
This study will explore what effects, if any, direct current (DC) brain polarization may produce on mental processes, such as attention, reaction time, working memory, speed of information processing and mood or emotional states. In DC brain polarization, a very weak electrical current is applied to the head. This technique has been used for many years on patients and healthy people with no known serious side effects. Studies have shown that DC polarization can temporarily improve people's ability to think of certain words. To determine if DC polarization can be used as a treatment for certain types of brain disorders, its possible effects on mood and other mental abilities must be determined.

Healthy normal volunteers over age 18 may be eligible for this study.

In each of three 1.5-hour sessions scheduled a day apart, participants complete the tasks listed below to determine the effects of polarization. For each session, electrodes are placed on the head, arm, and hand. One set of electrodes is for brain stimulation; the second set is used to measure the amount of skin moisture on the hand. The participants' tasks are to:

* Push a button on a keyboard when they see a specific item.
* Circle a number or make a mark on a line to indicate how much they feel a particular emotion or sensation at that time.
* Answer questions about themselves, or their opinions on certain topics.
* Look at several pictures and say how emotional they think they are.
* Read about an imaginary situation and say what they would do in that situation.
* Choose between decks of cards to try to win money.
* Compare the angles of lines.
* Identify smells, using a scratch and sniff test.
* At the end of the session, say how they are feeling.

Participants are called by phone on the day after each session to see how they are feeling.

DETAILED DESCRIPTION:
Objective: The principal objective is to establish the safety and feasibility of bilateral direct current (DC) polarization of the frontal lobes, which may be a useful modality for treatment of frontal lobe cognitive or behavioral deficits. Our secondary objective is to gather preliminary data on whether DC can modulate cognitive and emotion-related functions of the frontal lobes in healthy individuals. Study population: 25 healthy volunteers between the ages of 18 and 80 will be enrolled. Design: The study is a double-blind crossover study with three arms: anodal polarization, cathodal polarization, and sham treatment. Outcome Measures: The primary outcome measures are 1) cognitive function as measured with the CalCAP battery or 2) emotional state as measured with the Profile of Mood States. Secondary outcome measures include tests of emotion-based decision making and social cognition.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers over age 18. Pregnant women are eligible.

EXCLUSION CRITERIA:

Presence of metal in the cranial cavity or any holes in the skull due to trauma or surgery.

Uncontrolled medical problems, such as diabetes mellitus, hypertension, airway disease, heart failure, coronary artery disease, or any other condition that poses a risk for the subject during participation.

Broken skin in the area of the electrodes.

Any history of a neurological or psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2007-01-11; Study Completion 2008-12-23

PRIMARY OUTCOMES:
Measure significant changes in psychomotor and cognitive function with the CalCAP battery or adverse changes in mood as measured by the Profile of Mood States.

SECONDARY OUTCOMES:
Screen for other cognitive, emotional, and perceptual changes using standardized and validated neuropsychological tests.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bechara A, Tranel D, Damasio H, Damasio AR. Failure to respond autonomically to anticipated future outcomes following damage to prefrontal cortex. Cereb Cortex. 1996 Mar-Apr;6(2):215-25. doi: 10.1093/cercor/6.2.215. PMID 8670652
- [Background] BINDMAN LJ, LIPPOLD OC, REDFEARN JW. Long-lasting changes in the level of the electrical activity of the cerebral cortex produced bypolarizing currents. Nature. 1962 Nov 10;196:584-5. doi: 10.1038/196584a0. No abstract available. PMID 13968314
- [Background] CREUTZFELDT OD, FROMM GH, KAPP H. Influence of transcortical d-c currents on cortical neuronal activity. Exp Neurol. 1962 Jun;5:436-52. doi: 10.1016/0014-4886(62)90056-0. No abstract available. PMID 13882165